CLINICAL TRIAL: NCT01452984
Title: Experience of Patients With Non-Melanoma Skin Cancer of the Head and Neck Undergoing Mohs Surgery
Brief Title: Experience of Non-Melanoma Skin Cancer (NMSC) Mohs Surgery Project
Status: Completed | Type: Observational
Sponsor: Abramson Cancer Center at Penn Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: UPCC 07311
Record Dates: First submitted 2011-10-13; First posted 2011-10-17 (Estimated); Last update posted 2015-03-19 (Estimated); Status verified 2015-03

CONDITIONS: Non-Melanoma Skin Cancer
Keywords: Non-Melanoma skin cancer patients who have undergone or about to undergo Mohs surgery; who are treated within the University of Pennsylvania Health System

STUDY DESIGN:
Observational Model: Cohort
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Single Retrospective Interviews: Each retrospective interview will be conducted by the Principal Investigator and/or Project Manager to collect denmographic information and experiential narratives from the patient, using open-ended questions and structured probes based on individual responses. Retrospective interviews will be recorded and scheduled at the patients' convenience either in the clinic, at the home, or at a place that is convenient to them.
- Prospective Observations: Prospective Observations of clinic visits will be combined with informal interview to document conversations with their treating physicians about concerns emerging from appearance, function, and other factors that may impinge on clinical decision making and experience including quality of life. The Project Manager will be present for the clinical visit during which the Mohs surgery takes place and record field observations as well as informal interview notes in a notebook.

SUMMARY:
Mohs surgery excises non-melanoma skin cancer tumors of the head and neck while preserving maximum healthy tissue, an advantageous characteristic when dealing with the cosmetic and functional cervifacial region. Yet, treatment can result in changes to function and appearance with effects on quality of life. This project uses Grounded Theory to explore the Mohs surgery experience of NMSC patients who have head and neck lesions through interview and observation of the surgical appointment.

DETAILED DESCRIPTION:
Mohs surgery offers significant benefits in excising NMSC tumors of the head and neck by precisely removing cancerous tissue while preserving the maximum amount of healthy tissue, a characteristic of particular advantage when dealing with NMSC in the highly cosmetic and functional cericofacial region. Despite this, few studies have explored the patient perspective on their experience with Mohs surgery. Futhermore, treatment for NMSC can result in scarring, disfigurement, and changes to function and appearance. Ramifications on identity and self, embodiment and aesthetics, interaction and relationships appear likely and consequences on function and quality of life might then follow. Using Grounded Theory, this project aims to explore the question "what is the experience of Mohs surgery for non-melanoma skin cancer patients who have lesions of the head and neck?" Potential patient participants are those diagnosed with non-melanoma skin cancer, who have undergone Mohs surgery or are scheduled to undergo Mohs surgery on skin located in any area above the shoulders, and are referred to the project by their surgeons. They will represent a range of disease, from those who have had a single Mohs surgery to those with recurrent NMSC and repeated Mohs. Patients will also read and speak English and be at least 18 years of age. Transcribed interviews and field notes will be analyzed using constant comparative technique to develop descriptive and theoretical understandings of how experience Mohs surgery for non-melanoma skin cancer of the head and nexk.

ELIGIBILITY:
Inclusion Criteria:

* Patient participants must have an upcoming Mohs surgery scheduled or have already undergone Mohs surgery within the University of Pennsylvania Health System.
* All participants must read and speak English.
* For those patient participants with communication impairments due to surgery and treatment, accomodations for alternate methods of communication, including typing responses to the interview guide into a laptop computer or writing responses with a pen on paper, will be provided.
* Both male and female
* Must read and speak English
* Be over the age 18 and able to give consent.

Exclusion Criteria:

* This study excludes patients and their partners who are incapacitated or not old enough to give consent, more specifically those under the age of 18.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: This study involves non-melanoma skin cancer patients who have undergone or are about to undergo Mohs surgery, who are treated within the University of Pennsylvania Health System.
Sampling Method: Non-Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2011-07; Primary Completion 2013-12 (Actual); Study Completion 2013-12 (Actual)

PRIMARY OUTCOMES:
Number of Adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Sarah Kagan, PhD, RN, Principal Investigator — Abramson Cancer Center at Penn Medicine
Locations (1):
- Abramson Cancer Center of the University of Pennsylvania, Philadelphia, Pennsylvania, United States